CLINICAL TRIAL: NCT04613258
Title: Soy, Catfish, Anchovy, and Rice Supplementation Increases 25(OH)D Serum Levels in Tuberculosis Patients With Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, DINA KEUMALA SARI, Principal Investigator, Universitas Sumatera Utara
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: USU
Record Dates: First submitted 2020-09-29; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Tuberculosis
Keywords: polymorphism; porridge; vitamin D; biomolecular
MeSH Terms: conditions — Tuberculosis | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: We aimed to determine the effect of soy, catfish, anchovy, and rice (SCAR) porridge supplementation for 14 days along with nutritional counseling on vitamin D, calcium, and biomolecular parameters on new patients diagnosed with tuberculosis and associated complications who visited two public health centers: Teladan Public Health Center and Amplas Public Health Center, located in Medan, North Sumatera, Indonesia. The sample was collected on Sumatera Island, at latitude 3.57 N and longitude 98.65 E, with enough sunlight and a temperature of ± 32 °C (90 °F). The study was performed from May to September 2019. This study was a controlled randomized clinical trial. After applying the inclusion and exclusion criteria, 43 patients participated in the study. These patients were divided into two groups: 22 patients were put into the treatment group (I) and 21 into the control group (C).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCAR Porridge Group (Active Comparator): There were 22 subjects in the intervention group (I) who received 50 g of SCAR porridge once per day, along with dietary counseling.
  Interventions: Dietary Supplement: SCAR Porridge
- Counseling Group (Active Comparator): 21 subjects in the control group (C) who only received dietary counseling
  Interventions: Other: Counseling

INTERVENTIONS:
Dietary Supplement: SCAR Porridge — The treatment group was given SCAR porridge supplementation in the form of a soft porridge (a mixture of 50 g dry powder porridge added to 200 mL of hot water) along with nutritional counseling. The control group only received nutritional counseling and no SCAR porridge supplementation. A 50 g portion of SCAR porridge was provided once a day for 14 days. The SCAR porridge was monitored and administered by a researcher once a week to inquire about adherence to the supplementation consumption and perceived side effects. All research subjects went through a clearance period of one week and were requested not to consume any supplements.
  Arms: SCAR Porridge Group
Other: Counseling — 21 subjects in the control group (C) who only received dietary counseling
  Arms: Counseling Group

SUMMARY:
Tuberculosis patients that have complications (e.g., diabetes mellitus and human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS)) who live in tropical regions experience vitamin D deficiency, especially in North Sumatra, Indonesia. The presence of vitamin D receptor (VDR) polymorphism genes, TaqI and FokI, is one of the predisposing factors, as is high levels of inflammatory markers, also indicating disease progression and malnutrition. This study aims to assess the effect of 50 g of soy-catfish-anchovy-rice (SCAR) porridge per day for 14 days on 25(OH)D, calcium, and biomolecular serum levels in patients with VDR gene polymorphisms (TaqI or FokI). The study was a parallel, open, clinical trial. A total of 43 subjects with the VDR gene polymorphisms were selected. The subjects were divided into two groups using block randomization. There were 22 subjects in the intervention group (I) who received 50 g of SCAR porridge once per day, along with dietary counseling, and 21 subjects in the control group (C) who only received dietary counseling.

DETAILED DESCRIPTION:
Tuberculosis patients that have complications (e.g., diabetes mellitus and human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS)) who live in tropical regions experience vitamin D deficiency, especially in North Sumatra, Indonesia. The presence of vitamin D receptor (VDR) polymorphism genes, TaqI and FokI, is one of the predisposing factors, as is high levels of inflammatory markers, also indicating disease progression and malnutrition. This study aims to assess the effect of 50 g of soy-catfish-anchovy-rice (SCAR) porridge per day for 14 days on 25(OH)D, calcium, and biomolecular serum levels in patients with VDR gene polymorphisms (TaqI or FokI). The study was a parallel, open, clinical trial. A total of 43 subjects with the VDR gene polymorphisms were selected. The subjects were divided into two groups using block randomization. There were 22 subjects in the intervention group (I) who received 50 g of SCAR porridge once per day, along with dietary counseling, and 21 subjects in the control group (C) who only received dietary counseling. All subjects in both groups completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants which have newly diagnosed with lung tuberculosis with an acid fast bacilli (AFB) result (+), aged 18-60 years, with a heterozygote genotype test performed on one of the genes TaqI and FokI, willing to participate in the study, and provided informed consent

Exclusion Criteria:

* Participants which being pregnant and/or a breastfeeding mother

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-05-11 (Actual); Primary Completion 2019-08-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Vitamin D | up to 2 weeks
  25(OH)D Serum level
Calcium | up to 2 weeks
  Calcium Serum level

SECONDARY OUTCOMES:
albumin | up to 2 weeks
  albumin serum level
Hs CRP | up to 2 weeks
  Hs CRP serum level
blood glucose | up to 2 weeks
  blood glucose serum level

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Universitas Sumatera Utara, Medan, North Sumatra, Indonesia

DOCUMENTS (2):
  • Informed Consent Form (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT04613258/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-05-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT04613258/Prot_SAP_001.pdf